CLINICAL TRIAL: NCT02115737
Title: Group Treatment for Adolescents With Depression
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Benjamin Goldstein, Associate Processor, University of Toronto, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 213-2012
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dialectical Behavior Therapy Skills Group (Experimental): Twelve week skills based group therapy include four modules: mindfulness, emotion regulation, distress tolerance, and walking the middle path
  Interventions: Behavioral: Dialectical Behavior Therapy Skills Group
- Psychoeducation group treatment (Experimental): The comparison group used in the present study is based on a publicly available treatment manual from the Services for Teens At Risk (STAR) Center at the University of Pittsburgh
  Interventions: Behavioral: Psychoeducation group treatment

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy Skills Group
  Arms: Dialectical Behavior Therapy Skills Group
Behavioral: Psychoeducation group treatment
  Arms: Psychoeducation group treatment

SUMMARY:
Youth with depressive symptoms are at risk for a range of problems later in life. This includes problematic interpersonal relationships, occupational stress, and the occurrence of adult mental disorders. The main purpose of this study is to test how effective two types of group therapy are at reducing depressive symptoms in youth. A focus on group therapy is important because group therapy allows for many youth to be treated in a short amount of time. Group therapy is also helpful because youth can get social support and feel less alone in their symptoms when they participate in group. This study compares two groups, one that targets skills for managing difficult emotional experiences (dialectical behavior therapy skills group) and another group focuses on psychoeducation and is based on a publicly available treatment manual from the Services for Teens At Risk (STAR) Center at the University of Pittsburgh. The results of this study will provide insights regarding the comparative efficacy of these two treatments, and regarding predictors of treatment response.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* male or female, ages 14 to 19, all races and ethnicities
* Current depression as assessed by an ALIFE - PSR score equal to or greater than 4
* Has a treating psychiatrist at Sunnybrook Health Sciences Centre

Exclusion Criteria:

* Current manic episode
* current psychosis

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Actual)
Dates: Start 2013-12; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Children's Depression Rating Scale - Revise (CDRS-R) | Change from baseline to endpoint (assessed at weeks 0, 12, 24)
  Measure mood symptom severity. Response is defined as greater than or equal to 50% reduction in CDRS-R score
The Longitudinal Interval Follow-up Evaluation for adolescents (A-LIFE) | Change from baseline to endpoint (assessed at weeks 0, 12 and 24)
  Used to track symptom severity, treatment (both psychosocial and psychotropic), self-injurious/suicidal behavior and psychosocial functioning over time.

SECONDARY OUTCOMES:
The Adverse Childhood Experiences | Assessed at baseline
  Used to measure adverse events that have happened up until the 18th year of life
The Children's Affective Lability Scale | Change from baseline to endpoint (assessed at weeks 0, 4, 12 and 24)
  Used to ascertain adolescent and parent reported affect regulation, during the preceding year or time since last assessment
The Stressful Life Events Schedule | Change from baseline to endpoint (assessed at weeks 0, 4, 12, and 24)
  Used to ascertain 80 adolescent and parent reported negative life events, during the preceding year or time since last assessment
The DBT Ways of Coping Checklist | Change from baseline to endpoint (assessed at weeks 0, 4, 12, and 24)
  This is a self-reported questionnaire used to assess adaptive and maladaptive ways to cope with negative emotions or problematic situations
The Life Problems Inventory | Change from baseline to endpoint (assessed at weeks 0, 4, 12, and 24)
  This is a self-reported questionnaire (adolescent-reported) used to assess emotion dysregulation in the adolescent.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin I Goldstein, MD, Principal Investigator — Sunnybrook Health Science Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada